CLINICAL TRIAL: NCT07401732
Title: Prediction of Dysphagia Severity and Diagnosis of Its Possible Causes in Rheumatoid Arthritis: A Cross-Sectional Study
Brief Title: Dysphagia in Rheumatoid Arthritis
Status: Not yet recruiting | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Aliaa Mamdouh Adelaziz Farag, Lecturer, Tanta University
Other Study IDs: 36264PR772/7/24
Record Dates: First submitted 2026-01-21; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis (RA
Keywords: Flexible Endoscopic Evaluations of Swallowing; Temporomandibular joint; Deglutition disorders; cricoarytenoid
MeSH Terms: conditions — Arthritis, Rheumatoid; Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Interventional Study Model: Single Group Assignment (rheumatoid arthritis patients)
  Interventions: Diagnostic Test: flexible fiberoptic pharyngolaryngoscopy

INTERVENTIONS:
Diagnostic Test: flexible fiberoptic pharyngolaryngoscopy — Flexible Endoscopic Evaluations of Swallowing (FEES) will be used to examine the nose, throat, and airway to diagnose possible causes of dysphagia. The dysphagia severity scale via FEES will be scored. It is a flexible process that may be applied to a variety of situations and objectives (named as flexible pharyngolaryngoscopy). Following the routine oropharyngeal examination, its versatility can enable it to be used as a laryngoscope for examining the larynx and adjacent regions.

SUMMARY:
The primary goal of this cross-sectional study is to assess risk factors/predictors for dysphagia severity in RA.

The secondary goals include demonstrating whether flexible fiberoptic pharyngolaryngoscopy can diagnose joint-affection-induced dysphagia in patients with rheumatoid arthritis (RA) and whether both oropharyngeal and esophageal dysphagia are present among these patients.

The main questions it aims to answer are

* What are the predictors that are associated with dysphagia severity via flexible fiberoptic pharyngolaryngoscopy in rheumatoid arthritis patients?
* Whether flexible fiberoptic pharyngolaryngoscopy can diagnose joint-affection-induced dysphagia in patients with RA?
* Whether both oropharyngeal and esophageal dysphagia are present in patients with RA?

DETAILED DESCRIPTION:
This cross-sectional study will comprise RA patients during their visits to inpatient and outpatient clinics. The inclusion criterion is patients with RA defined by the American College of Rheumatology/European League Against Rheumatism collaborative initiative (ACR/EULAR) 2010 classification criteria. Patients aged above 18 years old, well-orientated, and cooperative.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Rheumatoid arthritis defined by the American College of Rheumatology/European League Against Rheumatism collaborative initiative (ACR/EULAR) 2010 classification criteria.
* Patients aged above 18 years old, well-orientated, and cooperative.

Exclusion Criteria:

* concomitant cancer diagnosis, pregnancy.
* jaw-related traumas, teeth and gum diseases.
* other rheumatologic conditions
* other comorbidities.
* other causes of TMJ arthritis, patients with TMJ, palatal or tongue congenital abnormalities, and patients who underwent TMJ injections in the last six months.
* Patients with any language disorders or intellectually handicapped (as certain questions depend on the patient's ability to comprehend and express their emotions regarding their issue) and patients with anatomical anomalies impeding the functionality of flexible nasofibroscopy.
* Any apparent causes of dysphagia other than RA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with RA defined by the American College of Rheumatology/European League Against Rheumatism collaborative initiative (ACR/EULAR) 2010 classification criteria.
Sampling Method: Probability Sample
Enrollment: 137 (Estimated)
Dates: Start 2026-02-07 (Estimated); Primary Completion 2026-03-05 (Estimated); Study Completion 2026-03-05 (Estimated)

PRIMARY OUTCOMES:
Identifying potential predictors of dysphagia severity in rheumatoid arthritis patients. | The assessment of dysphagia severity via FEES typically will take nearly 25 minutes. The duration of clinical, laboratory, and radiological tests will take 1 to 2 days and may vary depending on the specific circumstances.
  Demonstrating the associations between the dysphagia severity scale (DSS) via flexible/fibre-optic endoscopic evaluations of swallowing (FEES) and the following:
  1. Active disease by disease activity score in 28 joints with C-reactive protein (DAS28-CRP ): low if DAS28-CRP score was less than 3.2, moderate if the score between 3.2 and 5.1, or high if the score > 5.1.
  2. RA patient's malfunction by Modified Health Assessment Questionnaire (MHAQ): mild functional loss if score less than 1.3, moderate if score between 1.3 and 1.8, severe loss if > 1.8
  3. Temporomandibular dysfunction: mild TMJ dysfunction if score from 20 to 40, moderate dysfunction if score from 45 to 65 and severe TMJ dysfunction if the score from 70 to 100.
  4. Increased serum thyroid-stimulating hormone (TSH) > 5 mU/L
  5. Erosion in temporomandibular (TMJ) and/or cricoarytenoid (CAJ) joints by cone beam CT imaging.

SECONDARY OUTCOMES:
Demonstrating whether flexible fiberoptic pharyngolaryngoscopy can diagnose Joint-Affection-Induced dysphagia in patients with RA. | Assessment of rheumatoid arthritis patients by FEES will take 10 to 25 minutes. The duration may vary depending on the specific circumstances and the complexity of the assessment.
  Flexible Endoscopic Evaluations of Swallowing (FEES) will be used to examine the nose, throat, and airway to diagnose possible causes of dysphagia. It is a flexible process that may be applied to a variety of situations and objectives (named as flexible pharyngolaryngoscopy). Following the routine oropharyngeal examination, its versatility can enable it to be used as a laryngoscope for examining the larynx and adjacent regions.
Demonstrating whether both oropharyngeal and oesophageal dysphagia are present among patients with RA? | up to 2 minutes following routine FEES.
  An upper oesophagus examination by FEES may provide a useful screening tool for oesophageal dysphagia in addition to the routine oropharyngeal and laryngeal examination.

CONTACTS AND LOCATIONS:
Overall Officials: Aliaa MA Farag, MD, Principal Investigator — Tanta University Faculty of Medicine
Locations (1):
- Faculty of medicine, Tanta University, Tanta, Elgharbia, Egypt

IPD SHARING:
Plan to Share IPD: No
Data is available with corresponding author on reasonable request.